CLINICAL TRIAL: NCT05592847
Title: The Effect of a Nurse Navigator Program on Readmission Rates for Patients With Elevated BMI, COPD, CHF, Dialysis Use, and H/o Alcohol Abuse
Brief Title: A Study of the Effect of a Nurse Navigator Program on High Risk Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, George Pujalte, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-013158
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Patient Readmission; Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip; Heart Failure; Pulmonary Disease, Chronic Obstructive; Renal Insufficiency; Body Mass Index; Alcoholism
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Renal Insufficiency; Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Practice (No Intervention): Patients with chronic conditions slated for surgery contacted once by pre-operative nurse to discuss surgery
- Nurse Navigator (Experimental): Patients with chronic conditions slated for surgery contacted once by pre-operative nurse to discuss surgery, then contacted at intervals by nurse navigator study team members
  Interventions: Other: Nurse Navigator Program

INTERVENTIONS:
Other: Nurse Navigator Program — Identification of specific chronic conditions and suggestion of management care of primary care physicians and referrals to specialists via nurse navigator team members.
  Arms: Nurse Navigator

SUMMARY:
The purpose of this study is to examine if educational intervention in high risk patients can lead to decreased hospital readmissions when compared to patients who are not in the intervention program. Additionally, to determine patient satisfaction with the educational program.

ELIGIBILITY:
Inclusion Criteria:

- Require total or partial hip or knee replacement and have one or more of the following diagnosis: Heart Failure (HF); Chronic obstructive pulmonary disease (COPD); Dialysis; Alcohol Abuse; Low BMI.

Exclusion Criteria:

- Decrease cognitive capacity to consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Readmission rates | One year

CONTACTS AND LOCATIONS:
Overall Officials: George Pujalte, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials